CLINICAL TRIAL: NCT07276802
Title: The TRIBECA Study (TRIessence/Byqlovi for Easier CAtaract Surgery)
Acronym: TRIBECA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 250501 TRIBECA
Record Dates: First submitted 2025-10-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-10

CONDITIONS: Post Cataract Surgery
Keywords: Interventional Study Design
MeSH Terms: interventions — Triamcinolone; Clobetasol; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Group (Experimental): Triesence or Byqlovi Arm with nepafenac
  Interventions: Drug: Triamcinolone (Optional)
- Control Group (Active Comparator): Topical Moxifloxacin, Ketorolac, Prednisolone Acetate
  Interventions: Drug: control group

INTERVENTIONS:
Drug: Triamcinolone (Optional) — triamcinolone 40mg/ml or topical clobetasol 0.05% with nepafenac 0.3% QD for 14 days
  Other Names: clobetasol
  Arms: Experimental Group
Drug: control group — topical medication regimen will include prednisolone acetate 1% QID, ketorolac 0.5% QID, and moxifloxacin 0.5% topical drops QID.
  Arms: Control Group

SUMMARY:
A self-controlled, prospective clinical study of the safety, clinical efficacy, and patient acceptance of subconjunctival delivery of triamcinolone 40 mg/mL (Triesence) at the conclusion of cataract surgery or topical clobetasol 0.05 (Byqlovi) BID for 14 days, with intracameral moxifloxacin 0.5%, and topical nepafenac 0.3% (Ilevro) for 14 days, as compared to traditional topical postoperative prednisolone acetate 1% QID, moxifloxacin 0.5% drops QID, and ketorolac 0.5% QID in controlling postoperative pain and inflammation in subjects undergoing sequential bilateral cataract surgery.

DETAILED DESCRIPTION:
Drug delivery is one of the most exciting advances in ophthalmology, and with new products available comes the opportunity for an improved patient experience in cataract surgery. Frequent use of topical medications is associated with difficulty in application and compliance for many patients and create a burden for family members. In addition there is a cost to many patients that presents financial obstacles.

The purpose of this study is to evaluate the safety, effectiveness and patient acceptance of two post cataract surgery drug treatment regimens that minimize the use of topical medications. This will be a prospective evaluation of patients having routine, bilateral cataract surgery in which one eye of each subject will be randomized to receive a "conventional" regimen and the other eye will receive a regimen of "less drops". The "less drops" regimen will include EITHER (by randomization) a 0.1 cc subconjunctival injection of triamcinolone 40mg/mL (Triesence) at the end of surgery OR postoperative administration of topical clobetasol 0.05% (Byqlovi) BID for 14 days to deliver corticosteroid. Both steroid regimens will be delivered with nepafenac 0.3% QD for 14 days as a topical NSAID, and intracameral moxifloxacin 0.5% QID for 7 days as an antibiotic. The "conventional" topical medication regimen will include prednisolone acetate 1% QID, ketorolac 0.5% QID , and moxifloxacin 0.5% topical drops QID. With all of these treatment regimens, the patients will be receiving two on-label, FDA approved products and one (intracameral moxifloxacin) that is technically off-label but is so well accepted that it is used in approximately half the cataract surgery performed in the US. . In all patients the fellow eye will act as the control.

Patients will be evaluated at 1 day, 1 week and 1 month postoperatively. Measurements are listed in the visit schedule table below. Patients will also be subjectively asked about their symptoms of pain and photophobia and be asked about their acceptance, cost, and which treatment protocol they preferred.

ELIGIBILITY:
Inclusion Criteria:

* A male or female subject in good general health, > 22 years of age at the time of the screening visit
* A subject must be able to comprehend and willing to give informed consent
* A woman of child-bearing potential must not be pregnant or lactating.
* A subject has the availability, willingness and sufficient cognitive awareness to comply with exam procedures and able to return for all scheduled study visits
* A subject with a cataract for which routine phacoemulsification extraction and implantation of an intraocular lens has been planned
* A subject with clear ocular media other than cataract in their scheduled operative eye
* A subject with normal OCT of the macula in both eyes
* A subject has the potential for a post-operative Snellen BCDVA of 20/30 or better in both eyes

Exclusion Criteria:

* A subject with a history of complications, adverse events, trauma or disease in the nasolacrimal area, whether or not it was due to punctal plug wear, including but not limited to dacryocystitis, inflammation or canaliculitis in either eye
* A subject with any moderate to severe lid, conjunctival or corneal findings in either eye at the screening visit
* A subject with any signs of intraocular inflammation (cells/flare) in either eye at the screening visit
* A subject with a known sensitivity to any of the study medications.
* A subject with a history as a steroid responder or glaucoma
* A subject with a known or suspected allergy or hypersensitivity to non-steroidal anti-inflammatory drugs (NSAIDs), or to any component of the test article
* A subject with only one eye with potentially good vision
* A subject with a known pathology that may affect visual acuity (as determined by the Investigator); particularly retinal changes that affect vision (macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, etc.) in their scheduled surgical eye
* A subject that has a condition associated with the fluctuation of hormones that could lead to refractive changes
* A subject with amblyopia or strabismus
* A subject has a history of ocular trauma in their scheduled surgical eye
* A subject that has undergone prior intraocular surgery in the scheduled surgical eye within the last 6 months or laser surgery within three months prior to screening
* A subject with pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 3.5 mm under mesopic/scotopic conditions) in their scheduled surgical eye.
* A subject with a clinically significant corneal abnormality (e.g., stromal, epithelial or endothelial dystrophies) that, in the best judgment of the investigator, is likely to interfere with the outcomes of the study
* A subject with an inability to achieve keratometric stability for contact lens wearers
* A subject with a history of chronic/recurrent inflammatory eye disease (e.g., scleritis, uveitis, herpes keratitis) in either eye
* A subject with uncontrolled glaucoma
* A subject that requires the use of systemic or ocular medications that may affect vision, ocular inflammation or pain
* A subject with an acute or chronic disease, or illness, that would increase risk or confound study results (e.g., autoimmune disease, connective tissue disease, immunocompromised, suspected glaucoma, glaucomatous changes in the fundus or visual field, other source of ocular inflammation, etc.)
* A subject with an uncontrolled systemic disease: A potential subject in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study
* A subject with diabetes that is poorly controlled
* A subject currently participating or has participated in another clinical trial within 30 days prior to enrollment.

Intra-Operative Exclusion Criteria (Surgical Complications):

* Sulcus-sulcus or bag-sulcus fixation
* Posterior capsular rupture or zonular dialysis
* Disruption of anterior hyaloid face
* Vitreous loss
* Floppy iris syndrome
* Inability to place IOL in capsular bag
* Significant anterior chamber hyphema
* Significant zonular rupture.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary | 14 days after cataract surgery in each eye
  Patient Preference Between Medication Protocols (COMTOL Questionnaire Question 1)
Primary | 14 days after cataract surgery in each eye
  Patient preference for medication protocol between the two eyes, as reported based on the question, "Thinking about your overall experience taking medications in each eye after surgery, which eye did you prefer?" (question 1 from validated COMTOL questionnaire)

SECONDARY OUTCOMES:
Patient-Reported Postoperative Ocular Pain Severity Using a 0-10 Visual Analog Scale | 14 days after cataract surgery in each eye
  Study subject evaluation of post-op ocular pain using a visual analog scale with pain ranking from 0 to 10 (10 high) with the request, "Please rate the severity of discomfort caused by your eye medicines at their worst point."

OTHER OUTCOMES:
Summed Ocular Inflammation Score at One Week (Anterior Chamber Cells + Flare) | 7 days after cataract surgery in each eye
  Summed Ocular Inflammation Score (sum of the mean anterior chamber cells and anterior flare score) at one week.

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard Eye Associates, Laguna Hills, California, United States